CLINICAL TRIAL: NCT00790205
Title: TECOS: A Randomized, Placebo Controlled Clinical Trial to Evaluate Cardiovascular Outcomes After Treatment With Sitagliptin in Patients With Type 2 Diabetes Mellitus and Inadequate Glycemic Control
Brief Title: Sitagliptin Cardiovascular Outcomes Study (MK-0431-082)
Acronym: TECOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Duke Clinical Research Institute, Oxford Diabetes Trials Unit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-082; 2008_523 (Other: Merck study number); 2008-006719-20 (EudraCT Number)
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin tablet taken orally once daily in the morning for up to approximately 5 years.
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Placebo to sitagliptin tablet taken orally once daily in the morning for up to approximately 5 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin, one 50 mg or one 100 mg tablet (dose dependant on renal function) orally, once daily.
  Other Names: MK-0431; Januvia®
  Arms: Sitagliptin
Drug: Placebo — Placebo tablet matching the 50 mg or 100 mg sitagliptin tablet, orally, once daily.
  Arms: Placebo

SUMMARY:
This is a clinical trial designed to assess the cardiovascular outcome of long-term treatment with sitagliptin used as part of usual care compared to usual care without sitagliptin in participants with type 2 diabetes mellitus (T2DM) having a history of cardiovascular (CV) disease and a hemoglobin A1c (HbA1c) of 6.5% to 8.0%.

Primary hypothesis A is that sitagliptin, when used as part of usual care, is non-inferior to usual care without sitagliptin with regard to the risk of developing a confirmed event in the primary CV composite endpoint of Major Adverse Cardiovascular Event (MACE) plus. If hypothesis A is satisfied: hypothesis B is that sitagliptin, when used as part of usual care, is superior to usual care without sitagliptin with regard to the risk of developing a confirmed event in the primary CV composite endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Has T2DM
* Has HbA1c between 6.5% (48 mmol/mol) and 8.0% (64 mmol/mol) on stable dose(s) of antihyperglycemic agent(s), including insulin
* Has pre-existing cardiovascular disease

Exclusion Criteria:

* Has a history of type 1 diabetes mellitus or ketoacidosis.
* Is not able to take sitagliptin

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14671 (Actual)
Dates: Start 2008-12-10 (Actual); Primary Completion 2015-03-30 (Actual); Study Completion 2015-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Green JB, Bethel MA, Paul SK, Ring A, Kaufman KD, Shapiro DR, Califf RM, Holman RR. Rationale, design, and organization of a randomized, controlled Trial Evaluating Cardiovascular Outcomes with Sitagliptin (TECOS) in patients with type 2 diabetes and established cardiovascular disease. Am Heart J. 2013 Dec;166(6):983-989.e7. doi: 10.1016/j.ahj.2013.09.003. Epub 2013 Oct 23. PMID 24268212
- [Result] Bethel MA, Green JB, Milton J, Tajar A, Engel SS, Califf RM, Holman RR; TECOS Executive Committee. Regional, age and sex differences in baseline characteristics of patients enrolled in the Trial Evaluating Cardiovascular Outcomes with Sitagliptin (TECOS). Diabetes Obes Metab. 2015 Apr;17(4):395-402. doi: 10.1111/dom.12441. Epub 2015 Feb 13. PMID 25600421
- [Result] Green JB, Bethel MA, Armstrong PW, Buse JB, Engel SS, Garg J, Josse R, Kaufman KD, Koglin J, Korn S, Lachin JM, McGuire DK, Pencina MJ, Standl E, Stein PP, Suryawanshi S, Van de Werf F, Peterson ED, Holman RR; TECOS Study Group. Effect of Sitagliptin on Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2015 Jul 16;373(3):232-42. doi: 10.1056/NEJMoa1501352. Epub 2015 Jun 8. PMID 26052984
- [Derived] Gao N, Dakin HA, Holman RR, Lim LL, Leal J, Clarke P. Estimating Risk Factor Time Paths Among People with Type 2 Diabetes and QALY Gains from Risk Factor Management. Pharmacoeconomics. 2024 Sep;42(9):1017-1028. doi: 10.1007/s40273-024-01398-4. Epub 2024 Jun 26. PMID 38922488
- [Derived] Bethel MA, Sourij H, Stevens SR, Hannan K, Lokhnygina Y, Adler AI, Peterson ED, Holman RR, Lopes RD. Time-dependent event accumulation in a cardiovascular outcome trial of patients with type 2 diabetes and established atherosclerotic cardiovascular disease. Cardiovasc Diabetol. 2023 Mar 28;22(1):72. doi: 10.1186/s12933-023-01802-x. PMID 36978066
- [Derived] Sharma A, Zheng Y, Ezekowitz JA, Westerhout CM, Udell JA, Goodman SG, Armstrong PW, Buse JB, Green JB, Josse RG, Kaufman KD, McGuire DK, Ambrosio G, Chuang LM, Lopes RD, Peterson ED, Holman RR. Cluster Analysis of Cardiovascular Phenotypes in Patients With Type 2 Diabetes and Established Atherosclerotic Cardiovascular Disease: A Potential Approach to Precision Medicine. Diabetes Care. 2022 Jan 1;45(1):204-212. doi: 10.2337/dc20-2806. PMID 34716214
- [Derived] McAlister FA, Zheng Y, Westerhout CM, Buse JB, Standl E, McGuire DK, Van de Werf F, Green JB, Armstrong PW, Holman RR; TECOS Study Group. Association between glycated haemoglobin levels and cardiovascular outcomes in patients with type 2 diabetes and cardiovascular disease: a secondary analysis of the TECOS randomized clinical trial. Eur J Heart Fail. 2020 Nov;22(11):2026-2034. doi: 10.1002/ejhf.1958. Epub 2020 Jul 28. PMID 32621557
- [Derived] De Ferrari GM, Stevens SR, Ambrosio G, Leonardi S, Armstrong PW, Green JB, Wamil M, Holman RR, Peterson ED; TECOS Study Group. Low-density lipoprotein cholesterol treatment and outcomes in patients with type 2 diabetes and established cardiovascular disease: Insights from TECOS. Am Heart J. 2020 Feb;220:82-88. doi: 10.1016/j.ahj.2019.11.005. Epub 2019 Nov 13. PMID 31790905
- [Derived] Shavadia JS, Zheng Y, Green JB, Armstrong PW, Westerhout CM, McGuire DK, Cornel JH, Holman RR, Peterson ED. Associations between beta-blocker therapy and cardiovascular outcomes in patients with diabetes and established cardiovascular disease. Am Heart J. 2019 Dec;218:92-99. doi: 10.1016/j.ahj.2019.09.013. Epub 2019 Oct 20. PMID 31715435
- [Derived] Nauck MA, McGuire DK, Pieper KS, Lokhnygina Y, Strandberg TE, Riefflin A, Delibasi T, Peterson ED, White HD, Scott R, Holman RR. Sitagliptin does not reduce the risk of cardiovascular death or hospitalization for heart failure following myocardial infarction in patients with diabetes: observations from TECOS. Cardiovasc Diabetol. 2019 Sep 3;18(1):116. doi: 10.1186/s12933-019-0921-2. PMID 31481069
- [Derived] Guimaraes PO, Peterson ED, Stevens SR, Lokhnygina Y, Green JB, McGuire DK, Holman RR, Lopes RD. Antithrombotic treatment gap among patients with atrial fibrillation and type 2 diabetes. Int J Cardiol. 2019 Aug 15;289:58-62. doi: 10.1016/j.ijcard.2019.04.085. Epub 2019 Apr 30. PMID 31079973
- [Derived] Reed SD, Li Y, Leal J, Radican L, Adler AI, Alfredsson J, Buse JB, Green JB, Kaufman KD, Riefflin A, Van de Werf F, Peterson ED, Gray AM, Holman RR; TECOS Study Group. Longitudinal medical resources and costs among type 2 diabetes patients participating in the Trial Evaluating Cardiovascular Outcomes with Sitagliptin (TECOS). Diabetes Obes Metab. 2018 Jul;20(7):1732-1739. doi: 10.1111/dom.13292. Epub 2018 Apr 20. PMID 29573215
- [Derived] Standl E, Stevens SR, Armstrong PW, Buse JB, Chan JCN, Green JB, Lachin JM, Scheen A, Travert F, Van de Werf F, Peterson ED, Holman RR; TECOS Study Group. Increased Risk of Severe Hypoglycemic Events Before and After Cardiovascular Outcomes in TECOS Suggests an At-Risk Type 2 Diabetes Frail Patient Phenotype. Diabetes Care. 2018 Mar;41(3):596-603. doi: 10.2337/dc17-1778. Epub 2018 Jan 8. PMID 29311155
- [Derived] Sharma A, Green JB, Dunning A, Lokhnygina Y, Al-Khatib SM, Lopes RD, Buse JB, Lachin JM, Van de Werf F, Armstrong PW, Kaufman KD, Standl E, Chan JCN, Distiller LA, Scott R, Peterson ED, Holman RR; TECOS Study Group. Causes of Death in a Contemporary Cohort of Patients With Type 2 Diabetes and Atherosclerotic Cardiovascular Disease: Insights From the TECOS Trial. Diabetes Care. 2017 Dec;40(12):1763-1770. doi: 10.2337/dc17-1091. Epub 2017 Oct 6. PMID 28986504
- [Derived] Pagidipati NJ, Navar AM, Pieper KS, Green JB, Bethel MA, Armstrong PW, Josse RG, McGuire DK, Lokhnygina Y, Cornel JH, Halvorsen S, Strandberg TE, Delibasi T, Holman RR, Peterson ED; TECOS Study Group. Secondary Prevention of Cardiovascular Disease in Patients With Type 2 Diabetes Mellitus: International Insights From the TECOS Trial (Trial Evaluating Cardiovascular Outcomes With Sitagliptin). Circulation. 2017 Sep 26;136(13):1193-1203. doi: 10.1161/CIRCULATIONAHA.117.027252. Epub 2017 Jun 16. PMID 28626088
- [Derived] Bethel MA, Engel SS, Green JB, Huang Z, Josse RG, Kaufman KD, Standl E, Suryawanshi S, Van de Werf F, McGuire DK, Peterson ED, Holman RR; TECOS Study Group. Assessing the Safety of Sitagliptin in Older Participants in the Trial Evaluating Cardiovascular Outcomes with Sitagliptin (TECOS). Diabetes Care. 2017 Apr;40(4):494-501. doi: 10.2337/dc16-1135. Epub 2017 Jan 5. PMID 28057693
- [Derived] Cornel JH, Bakris GL, Stevens SR, Alvarsson M, Bax WA, Chuang LM, Engel SS, Lopes RD, McGuire DK, Riefflin A, Rodbard HW, Sinay I, Tankova T, Wainstein J, Peterson ED, Holman RR; TECOS Study Group. Effect of Sitagliptin on Kidney Function and Respective Cardiovascular Outcomes in Type 2 Diabetes: Outcomes From TECOS. Diabetes Care. 2016 Dec;39(12):2304-2310. doi: 10.2337/dc16-1415. Epub 2016 Oct 14. PMID 27742728
- [Derived] Buse JB, Bethel MA, Green JB, Stevens SR, Lokhnygina Y, Aschner P, Grado CR, Tankova T, Wainstein J, Josse R, Lachin JM, Engel SS, Patel K, Peterson ED, Holman RR; TECOS Study Group. Pancreatic Safety of Sitagliptin in the TECOS Study. Diabetes Care. 2017 Feb;40(2):164-170. doi: 10.2337/dc15-2780. Epub 2016 Sep 14. PMID 27630212
- [Derived] McGuire DK, Van de Werf F, Armstrong PW, Standl E, Koglin J, Green JB, Bethel MA, Cornel JH, Lopes RD, Halvorsen S, Ambrosio G, Buse JB, Josse RG, Lachin JM, Pencina MJ, Garg J, Lokhnygina Y, Holman RR, Peterson ED; Trial Evaluating Cardiovascular Outcomes With Sitagliptin (TECOS) Study Group. Association Between Sitagliptin Use and Heart Failure Hospitalization and Related Outcomes in Type 2 Diabetes Mellitus: Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2016 May 1;1(2):126-35. doi: 10.1001/jamacardio.2016.0103. PMID 27437883

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 14,671 participants were randomized to treatment, provided consent and did not have any Good Clinical Practice (GCP) deviations.
Groups:
- Placebo: Matching placebo tablet taken orally once daily in the morning for up to approximately 5 years
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 7332 | 7339
Treated | 7266 | 7274
Completed | 6972 | 6905
Not Completed | 360 | 434
Not completed — Lost to Follow-up | 61 | 71
Not completed — Withdrawal by Subject | 299 | 363

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 7332 | 7339 | 14671
Age, Customized [Number; unit: Participants] — Age is unknown for 320 participants
  Participants
    Adults 18 - 64 years | 3315 (7.9) | 3301 (8.0) | 65.5 (8.0)
    From 65 - 84 years | 3813 | 3821 | 7634
    85 years and over | 46 | 55 | 101
    Unknown age | 158 | 162 | 320
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2134 | 2163 | 4297
  Male | 5198 | 5176 | 10374
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Sitagliptin, n= 7254; Placebo, n= 7274; Total, n=14528
  mL/min/1.73 m^2 | 74.9 (21.3) | 74.9 (20.9) | 74.9 (21.1)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — Sitagliptin, n= 7330; Placebo, n= 7336; Total, n= 14666
  Percentage of HbA1c | 7.2 (0.5) | 7.2 (0.5) | 7.2 (0.5)
Urine albumin creatinine ratio [Mean (Standard Deviation); unit: g/mol Creatinine] — Sitagliptin, n= 2606; Placebo, n= 2542; Total, n= 5148
  g/mol Creatinine | 8.6 (37.4) | 8.4 (36.0) | 8.5 (36.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With First Confirmed Cardiovascular (CV) Event of Major Adverse Cardiovascular Event (MACE) Plus (Per Protocol Population)
Description: Primary composite CV endpoint of MACE plus which includes CV-related death, nonfatal MI, nonfatal stroke, or unstable angina requiring hospitalization.
Time Frame: Up to 5 years
Population: Per protocol population included all randomized participants who received study medication except those participants who did not contribute at least 1 day of data to the study analysis due to a major protocol violation that excluded all of their data.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7257 | 7266
Percentage of participants | 9.6 | 9.6
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Non-Inferiority or Equivalence — Hazard Ratio of Sitagliptin/Placebo: the between-treatment difference in time to the first primary composite CV outcome measure was assessed by the hazard ratio between the sitagliptin and placebo groups. The confidence interval for the hazard ratio was computed and compared to 1.30, the non-inferiority margin; p < 0.001, Cox proportional hazards model; Model stratified by region with treatment group only as explanatory variable; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.88 to 1.09]

2. Primary Outcome: Percentage of Participants With First Confirmed CV Event of Major Adverse Cardiovascular Event (MACE) Plus (Intent to Treat Population)
Description: as for outcome 1
Time Frame: Up to 5 years
Population: Intent to treat population included all randomized participants who received study medication, provided consent, and did not have a major GCP deviation.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7332 | 7339
Percentage of participants | 11.4 | 11.6
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Cox proportional hazards model; Model stratified by region with treatment group only as explanatory variable; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.89 to 1.08]

3. Secondary Outcome: Percentage of Participants With First Confirmed CV Event of MACE (Per Protocol Population)
Description: CV composite endpoint of MACE which includes CV-related death, nonfatal MI, or nonfatal stroke.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7257 | 7266
Percentage of participants | 8.4 | 8.3
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Cox proportional hazards model; Model stratified by region with treatment group only as explanatory variable; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.89 to 1.11]

4. Secondary Outcome: Percentage of Participants With First Confirmed CV Event of MACE (Intent to Treat Population)
Description: CV composite endpoint of MACE which includes CV-related death, nonfatal MI, or nonfatal stroke.
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7332 | 7339
Percentage of participants | 10.2 | 10.2
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, Cox proportional hazards model; Model stratified by region with treatment group only as explanatory variable; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.89 to 1.10]

5. Secondary Outcome: Percent Incidence of All-cause Mortality (Per Protocol Population)
Description: Percent incidence of all-cause mortality is reported as the percentage of participants who died due to any cause.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7257 | 7266
Percentage of participants | 4.7 | 4.3
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Hazard Ratio of Sitagliptin/Placebo: The between-treatment difference in mortality due to all causes was assessed by the hazard ratio between the Sitagliptin and Placebo groups; Test type: Superiority or Other; p = 0.435, Cox proportional hazards model; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.91 to 1.24]

6. Secondary Outcome: Percent Incidence of All-cause Mortality (Intent to Treat Population)
Description: Percent incidence of all-cause mortality is reported as the percentage of participants who died due to any cause.
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7332 | 7339
Percentage of participants | 7.5 | 7.3
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.875, Cox proportional hazards model; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.90 to 1.14]

7. Secondary Outcome: Percent Incidence of Congestive Heart Failure (CHF) Requiring Hospitalization (Per Protocol Population)
Description: Percent incidence of CHF requiring hospitalization was reported as the percentage of participants who were admitted to the hospital for CHF.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7257 | 7266
Percentage of participants | 2.8 [1.00 to 1.53] | 2.8 [0.84 to 1.33]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Hazard Ratio of Sitagliptin/Placebo: The between-treatment difference in CHF cases requiring hospitalization was assessed by the hazard ratio between the Sitagliptin and Placebo groups; Test type: Superiority or Other; p = 0.858, Cox proportional hazards model; Model stratified by region with treatment group and history of CHF at baseline as explanatory variables; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.81 to 1.19]

8. Secondary Outcome: Percent Incidence of CHF Requiring Hospitalization (Intent to Treat Population)
Description: as for outcome 7
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7332 | 7339
Percentage of participants | 3.1 [1.00 to 1.53] | 3.1 [0.84 to 1.33]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.983, Cox proportional hazards model; Model stratified by region with treatment group and history of CHF at baseline as explanatory variables; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.83 to 1.20]

9. Secondary Outcome: Change From Baseline in Renal Function Over Time (Per Protocol Population)
Description: Change in renal function based on estimated glomerular filtration rate [eGFR] using the Modification of Diet in Renal Disease [MDRD] method.
Time Frame: Baseline and up to 5 years
Population: Per protocol population included all randomized participants who received study medication except those participants who did not contribute at least 1 day of data to the study analysis due to a major protocol violation that excluded all of their data. Number of participants analyzed consists of those participants with a baseline value.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7182 | 7203
mL/min/1.73 m^2
  Month 4; Sitagliptin, n= 3859; Placebo, n= 3864 | -1.9 (14.2) | -0.8 (14.3)
  Month 8; Sitagliptin, n= 3562; Placebo, n= 3501 | -2.5 (14.9) | -0.9 (15.1)
  Month 12; Sitagliptin, n=4912, Placebo, n=4778 | -1.8 (15.8) | -0.5 (16.2)
  Month 24; Sitagliptin, n=4782, Placebo, n=4637 | -3.1 (17.9) | -1.7 (17.5)
  Month 36; Sitagliptin, n=2776, Placebo, n=2614 | -3.7 (18.0) | -1.6 (18.8)
  Month 48; Sitagliptin, n=1096, Placebo, n=1056 | -3.7 (18.3) | -2.8 (18.4)
  Month 60; Sitagliptin, n=79, Placebo, n=88 | -3.5 (18.2) | -6.4 (17.3)

10. Secondary Outcome: Change From Baseline in Renal Function Over Time (Intent to Treat Population)
Description: Change in renal function based on eGFR using the MDRD method.
Time Frame: Baseline and up to 5 years
Population: Intent to treat population included all randomized participants who received study medication, provided consent, and did not have a major GCP deviation. Number of participants analyzed consists of those participants with a baseline value.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7254 | 7274
mL/min/1.73 m^2
  Month 4; Sitagliptin, n=3949; Placebo, n=3977 | -1.8 (14.3) | -0.8 (14.3)
  Month 8; Sitagliptin, n=3687; Placebo, n=3648 | -2.4 (14.8) | -0.9 (15.2)
  Month 12; Sitagliptin, n=5082; Placebo, n=5015 | -1.8 (15.8) | -0.5 (16.3)
  Month 24; Sitagliptin, n=5157; Placebo, n=5071 | -3.2 (17.9) | -1.7 (17.7)
  Month 36; Sitagliptin, n=3037; Placebo, n=2942 | -3.8 (18.1) | -1.6 (18.7)
  Month 48; Sitagliptin, n=1237; Placebo, n=1210 | -4.0 (18.4) | -2.8 (18.3)
  Month 60; Sitagliptin, n=93; Placebo, n=106 | -4.2 (17.4) | -5.7 (17.2)

11. Secondary Outcome: Change From Baseline in HbA1c Over Time (Per Protocol Population)
Description: HbA1c is a measure of the percentage of glycated hemoglobin in the blood. Estimated mean difference between sitagliptin and placebo controlling for baseline HbA1c and region.
Time Frame: Baseline and up to 4 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7250 | 7258
Percentage of HbA1c
  Month 4; Sitagliptin, n=6632, Placebo, n=6588 | -0.3 (0.8) | 0.1 (0.9)
  Month 8; Sitagliptin, n=6294, Placebo, n=6197 | -0.3 (0.9) | 0.1 (1.0)
  Month 12; Sitagliptin, n=6217, Placebo, n=6092 | -0.2 (1.0) | 0.1 (1.0)
  Month 24; Sitagliptin, n=5668, Placebo, n=5475 | -0.1 (1.0) | 0.2 (1.1)
  Month 36; Sitagliptin, n=3227, Placebo, n=3083 | -0.1 (1.1) | 0.1 (1.1)
  Month 48; Sitagliptin, n=1271, Placebo, n=1224 | 0.0 (1.1) | 0.1 (1.2)
  Month 60; Sitagliptin, n=106, Placebo, n=108 | -0.1 (1.0) | 0.0 (0.9)

12. Secondary Outcome: Change From Baseline in HbA1c Over Time (Intent to Treat Population)
Description: as for outcome 11
Time Frame: Baseline and up to 4 years
Population: Intent to treat population included all randomized participants who received study medication, provided consent, and did not have a major GCP deviation. Number of participants analyzed consists of those participants in the intent to treat population with a baseline value.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7325 | 7331
Percentage of HbA1c
  Month 4: Sitagliptin, n= 6772; Placebo, n= 6738 | -0.3 (0.8) | 0.1 (0.9)
  Month 8: Sitagliptin, n= 6478; Placebo, n= 6414 | -0.2 (0.9) | 0.1 (1.0)
  Month 12: Sitagliptin, n= 6448; Placebo, n= 6384 | -0.2 (1.0) | 0.1 (1.0)
  Month 24: Sitagliptin, n= 6105; Placebo, n= 5975 | -0.1 (1.0) | 0.1 (1.1)
  Month 36: Sitagliptin, n= 3521; Placebo, n= 3439 | -0.1 (1.1) | 0.1 (1.1)
  Month 48: Sitagliptin, n= 1432; Placebo, n= 1383 | 0.0 (1.1) | 0.1 (1.2)
  Month 60: Sitagliptin, n= 123; Placebo, n= 128 | 0.0 (1.0) | 0.0 (1.0)

13. Secondary Outcome: Change From Baseline in Urine Albumin:Creatinine Ratio Over Time (Per Protocol Population)
Description: Change from baseline reflects the difference between the urine albumin:creatinine ratio reported time point and baseline value.
Time Frame: Baseline and up to 5 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: g/mol Creatinine
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 2590 | 2522
g/mol Creatinine
  Month 4; Sitagliptin, n=664; Placebo, n=688 | -2.2 (27.7) | -1.4 (24.6)
  Month 8; Sitagliptin, n=635; Placebo, n=597 | 1.7 (38.5) | 0.2 (45.3)
  Month 12; Sitagliptin, n=1126; Placebo, n=1059 | 0.8 (27.7) | 1.2 (33.1)
  Month 24; Sitagliptin, n=930; Placebo, n=892 | 0.7 (34.0) | 3.2 (31.6)
  Month 36; Sitagliptin, n=488; Placebo, n=513 | 2.5 (24.0) | 4.0 (31.0)
  Month 48; Sitagliptin, n=238; Placebo, n=233 | 1.3 (15.2) | 1.5 (25.5)
  Month 60; Sitagliptin, n=13; Placebo, n=17 | -2.7 (10.1) | 4.8 (15.4)

14. Secondary Outcome: Change From Baseline in Urine Albumin:Creatinine Ratio Over Time (Intent to Treat Population)
Description: as for outcome 13
Time Frame: Baseline and up to 5 years
Population: Intent to treat population included all randomized participants who received study medication, provided consent, and did not have a major GCP deviation. Number of participants analyzed consists of those participants in the intent to treat population with a baseline value for the outcome measure.
Measure: Mean (Standard Deviation); unit: g/mol Creatinine
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 2606 | 2542
g/mol Creatinine
  Month 4; n=677, n=713 | -2.1 (27.5) | -1.4 (24.1)
  Month 8; n=658, n=624 | 2.1 (39.4) | 0.5 (44.5)
  Month 12; n=1167, n=1115 | 1.3 (30.2) | 1.2 (32.3)
  Month 24; n=1011, n=964 | 0.5 (33.1) | 3.1 (30.7)
  Month 36; n=537, n=553 | 2.6 (25.8) | 3.9 (30.3)
  Month 48; n=265, n=256 | 1.9 (16.3) | 1.6 (24.5)
  Month 60; n=14, n=18 | -2.5 (9.7) | 6.4 (16.4)

15. Secondary Outcome: Percentage of Participants Who Initiated Chronic Insulin Therapy (Per Protocol Population)
Description: Chronic insulin therapy is defined as a continuous period of insulin use of more than 3 months.
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 5554 | 5601
Percentage of participants | 8.6 | 11.9
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, Cox proportional hazards model; Model stratified by region with treatment group only as explanatory variable; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.61 to 0.77]

16. Secondary Outcome: Percentage of Participants Who Initiated Chronic Insulin Therapy (Intent to Treat Population)
Description: Chronic insulin therapy is defined as a continuous period of insulin use of more than 3 months.
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 5608 | 5655
Percentage of participants | 9.7 | 13.2
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, Cox proportional hazards model; Model stratified by region with treatment group only as explanatory variable; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.63 to 0.79]

17. Secondary Outcome: Percentage of Participants With Initiation of Co-interventional Agent (Per Protocol Population)
Description: In participants not receiving insulin at baseline, time to addition of first co-interventional agent (i.e., next oral antihyperglycemic agent [AHA] or chronic insulin, where chronic insulin therapy is defined as a continuous period of insulin use of more than 3 months.)
Time Frame: Up to 5 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7257 | 7266
Percentage of participants | 18.9 | 24.5
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, Cox proportional hazards model; Model stratified by region with treatment group only as explanatory variable; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.65 to 0.75]

18. Secondary Outcome: Percentage of Participants With Initiation of Co-interventional Agent (Intent to Treat Population)
Description: In participants not receiving insulin at baseline, time to addition of first co-interventional agent (i.e., next oral AHA or chronic insulin, where chronic insulin therapy is defined as a continuous period of insulin use of more than 3 months.)
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 7332 | 7339
Percentage of participants | 21.7 | 27.9
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p < 0.001, Cox proportional hazards model; Model stratified by region with treatment group only as explanatory variable; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.68 to 0.77]

ADVERSE EVENTS:
Time Frame: Up to 68 months (including up to 28 days after last dose of study drug)
Description: All participants as treated (APaT) population includes participants who received at least one dose of study drug.
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 928/7266 | 909/7274
Other Adverse Events (participants affected / at risk) | 0/7266 | 0/7274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=7266) | Placebo (N=7274)
Anaemia (Blood and lymphatic system disorders) | 23 (24) | 23 (23)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 6 (6) | 6 (6)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pernicious anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hamartoma (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 2 (2) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Syringomyelia (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 2 (2)
Vertigo labyrinthine (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 1 (1)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Corneal degeneration (Eye disorders) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 1 (1) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (2) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Change of bowel habit (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (2)
Duodenal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 5 (5) | 3 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 3 (3) | 4 (4)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastritis (Gastrointestinal disorders) | 10 (10) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 (11) | 12 (14)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 (10) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 5 (5)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 12 (12) | 11 (12)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 6 (6) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 2 (2) | 1 (1)
Melaena (Gastrointestinal disorders) | 2 (2) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophageal food impaction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peptic ulcer perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 3 (3)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 8 (8) | 6 (8)
Small intestinal perforation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 6 (6)
Varices oesophageal (Gastrointestinal disorders) | 1 (2) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 3 (3) | 1 (1)
Asthenia (General disorders) | 2 (2) | 3 (3)
Chest pain (General disorders) | 6 (6) | 8 (8)
Device dislocation (General disorders) | 2 (2) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 0 (0)
Drug intolerance (General disorders) | 1 (1) | 0 (0)
Fat necrosis (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Granuloma (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal hyperaemia (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 17 (19) | 26 (31)
Puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Spinal pain (General disorders) | 1 (1) | 0 (0)
Submandibular mass (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic congestion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Corneal graft rejection (Immune system disorders) | 1 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Acute hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Appendicitis perforated (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (3) | 4 (4)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 6 (7) | 4 (4)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2)
Hepatitis C (Infections and infestations) | 3 (3) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex encephalitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Infected bites (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (2) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Mycetoma mycotic (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Scrub typhus (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 17 (17) | 19 (19)
Acetabulum fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chemical burns of eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 9 (9) | 9 (9)
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 7 (7) | 11 (11)
Fibula fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Humerus fracture (Injury, poisoning and procedural complications) | 4 (5) | 9 (9)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Patella fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprosthetic osteolysis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Prescribed overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Renal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Road traffic accident (Injury, poisoning and procedural complications) | 5 (6) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 5 (6) | 4 (5)
Splinter (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Testicular injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Tracheal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Urinary bladder rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Anticoagulation drug level increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (2)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 8 (8)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (9) | 5 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (9) | 21 (21)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Ankle impingement (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 8 (9) | 8 (8)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 13 (14) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 52 (54) | 35 (37)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 12 (12)
Adenocarcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Angioimmunoblastic T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (5)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 44 (50) | 55 (86)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15) | 10 (10)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 6 (6)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 14 (14)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 2 (2)
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 12 (12)
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 6 (7)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian granulosa-theca cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 7 (7)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6)
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pleomorphic liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 36 (36) | 45 (45)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 3 (3)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Retroperitoneal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (5)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 (38) | 38 (44)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 7 (7)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (13) | 20 (23)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
T-cell prolymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thymic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tongue cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tracheal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 7 (7)
Urethral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acoustic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Arachnoid cyst (Nervous system disorders) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 2 (2)
Basal ganglia haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 2 (2)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 1 (1)
Cervical cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 3 (3)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 2 (2) | 0 (0)
Complex partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 5 (5) | 6 (6)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 2 (2)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (3)
Epilepsy (Nervous system disorders) | 2 (3) | 3 (3)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 3 (3) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Monoplegia (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis crisis (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 2 (2)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Nerve root compression (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neurological symptom (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 2 (2) | 3 (3)
Partial seizures (Nervous system disorders) | 1 (1) | 3 (3)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Piriformis syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Postictal state (Nervous system disorders) | 1 (1) | 0 (0)
Radiculitis lumbosacral (Nervous system disorders) | 1 (1) | 0 (0)
Retrograde amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 4 (4)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord disorder (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Subdural effusion (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Thoracic outlet syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Ulnar tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo CNS origin (Nervous system disorders) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 3 (3)
Dissociative disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Drug dependence (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 2 (2) | 3 (4)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Nicotine dependence (Psychiatric disorders) | 1 (1) | 0 (0)
Paranoid personality disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 2 (2)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (2) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 6 (8) | 6 (6)
Calculus urinary (Renal and urinary disorders) | 2 (2) | 4 (4)
Haematuria (Renal and urinary disorders) | 6 (6) | 6 (6)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 10 (10) | 9 (11)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 4 (4) | 4 (5)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Stag horn calculus (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 4 (4)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 4 (4) | 6 (7)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 15 (15) | 11 (11)
Calculus prostatic (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epididymal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Orchitis noninfective (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatism (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 4 (4) | 3 (3)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 (18) | 30 (37)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 6 (9)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Angiodysplasia (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 6 (6) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Lymphorrhoea (Vascular disorders) | 1 (1) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study at least 30 days prior to submission for publication/presentation or at least 14 calendar days prior to submission for abstracts.